CLINICAL TRIAL: NCT04457050
Title: Insulin Resistance and Resistin In Non-Diabetic Patients With Chronic Hepatitis C Before and After Direct-Acting Antiviral Drugs.
Brief Title: Effect of Hepatitis C Clearance on Insulin Resistance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Sameh A. Lashen, Associate Professor of Internal Medicine., Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020966
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Insulin Resistance; Hepatitis C
MeSH Terms: conditions — Insulin Resistance; Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Non-Diabetic Hepatitis C infected patients (Experimental): 1. clinical examination,
  2. measurement of weight (Kg), height (meter), and waist circumference (cm).
  3. Calculation of the body mass index.
  4. Ultrasound abdominal examination.
  5. Laboratory Investigations including Complete blood count, Serum aspartate and alanine aminotransferases, serum albumin, serum bilirubin, serum gamma-glutamyl transpeptidase, and international normalization ratio. HCV-RNA quantification before treatment and 12 weeks after the end of therapy.. Serum lipid profile, fasting and post-prandial blood sugar, glycated hemoglobin A1c also included.
  6. Treatment of all patients with the available generic direct antivirals in Egypt (sofosbuvir/ledipasvir ± ribavirin or sofosbuvir plus daclatasvir ± ribavirin).
  7. Evaluation of insulin resistance using the homeostasis model assessment of insulin resistance before and 12 weeks after end of treatment.
  8. measurement of serum levels of resistin before and at 12 weeks after treatment.
  Interventions: Drug: Sofosbuvir 400 milligram; Drug: Daclatasvir 60 milligram; Drug: Ribavirin 400 milligram; Drug: Ledipasvir 90milligram/Sofosbuvir 400 milligram Tab

INTERVENTIONS:
Drug: Sofosbuvir 400 milligram — single daily dose of 400 milligrams
  Other Names: Soflanork 400 milligram; Gratisovir 400 milligram
Drug: Daclatasvir 60 milligram — single daily dose of 60 milligrams for 12 weeks
  Other Names: Daklanork 60 milligram; Daktavira 60 milligram
Drug: Ribavirin 400 milligram — weight based dose, 1200 mg for weight > 75 kilogram, and 1000 milligram if weight < 75 kilograms for 12 weeks
  Other Names: Riba 400 milligram
Drug: Ledipasvir 90milligram/Sofosbuvir 400 milligram Tab — single daily dose for 12 weeks
  Other Names: HARVONI; Soflanork plus

SUMMARY:
Chronic hepatitis C infection has been linked to insulin resistance, which is the essential component of metabolic syndrome and type 2 diabetes mellitus. Resistin; an adipokine, has been demonstrated to stimulate the secretion of several inflammatory factors known to play a role in the induction of insulin resistance. we investigated the changes in insulin resistance after hepatitis C clearance in the era of direct antivirals.

DETAILED DESCRIPTION:
the link between hepatitis C infection and insulin resistance has been established. Insuli resistance has been linked to poor response to interferon based therapy. recently, direct acting antiviral drugs are approved for hepatitis C elimination with high potency and safety. The aim of the study is to: 1. Determine the prevalence of insulin resistance among non-diabetic patients with chronic HCV infection. 2. Explore the impact of treatment with DAAs on insulin resistance among chronic HCV infected patients. 3. Investigate the role of insulin resistance as a potential prognostic factor for the response to DAAs. 4. Explore the utility of resistin as a potential biomarker IR among HCV infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C treatment-naïve;
* Non-diabetic patients.

Exclusion Criteria:

* Seropositivity for hepatitis B virus infection;
* Diabetes mellitus;
* Bbody mass index ≥ 30 Kg/M*2;
* History of alcohol consumption;
* Endocrinopathies that may affect the glycemic homeostasis;
* Other known causes of chronic liver disease; Hepatic decompensation [defined as history of gastrointestinal bleeding (melena and /or hematemesis), jaundice, coagulopathy, hepatic encephalopathy, and/or ascites]; bleeding diathesis;
* Connective tissue diseases;
* Autoimmune diseases;
* Cardiac, respiratory or renal disease.
* Patient receiving immuno-modulatory therapy or drugs that affect the blood glucose levels such as steroids or beta-blockers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change in the insulin resistance before and after hepatitis C clearance | at baseline and 12 weeks after sustained virologic response
  Assess the change in the value of Homeostatic Model Assessment for Insulin resistance (Homeostatic Model Assessment for Insulin Resistance) after hepatitis C treatment by calculating the HOMA-IR for all patients at baseline and the re-calculation at 12 weeks after viral clearance to clarify the impact of hepatitis C treatment by direct antiviral drugs on insulin sensitivity.

SECONDARY OUTCOMES:
Prevalence of insulin resistance among hepatitis C patients | at baseline
  Prevalence of insulin resistance among hepatitis C patients
Sustained virologic response | at 12 weeks after treatment
  Sustained virologic response

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No